CLINICAL TRIAL: NCT05465304
Title: Effect of Azithromycin on Pregnancy Prolongation in Women at Risk for Premature Labour
Brief Title: Effect of Azithromycin in Preventing Premature Labour
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Raghda R.S. Hussein, Assistant Professor of Clinical Pharmacy, Beni-Suef University
Other Study IDs: REC-H-PhBSU-21022
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pregnant With Complication
MeSH Terms: conditions — Pregnancy Complications | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: control group, included pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments (progesterone) for prolongation of pregnancy.
- Azithromycin group: the first test group, involved pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy plus azithromycin for 5 days every month
  Interventions: Drug: Azithromycin
- Azithromycin plus Clindamycin group: the second test group in which the pregnant women administerated Azithromycin and clindamycin (Dalacin®) vaginal gel 5 times per month.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — The assessment of efficacy of azithromycin in preventing premature labour.The duration between administrating azithromycin as monotherapy and polytherapy and labour is calculated
  Groups: Azithromycin group; Azithromycin plus Clindamycin group

SUMMARY:
This is a prospective observational case controlled study. The control group will include pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy.

The test group will involve pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy plus azithromycin

DETAILED DESCRIPTION:
A prospective randomized clinical study was conducted in the outpatient clinic of the gynecology department of Beni Suef University Hospital, Beni-Suef, Egypt, between October 01, 2021, and April 30, 2022. The study included 211 pregnant women aged between 20 to 41 years. These patients were randomized into three groups.

The first group which was the control group, included pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments (progesterone) for prolongation of pregnancy. While the second group which was the first test group, involved pregnant women, having intact membranes and are at risk of or in preterm labour, administrating the standard treatments for prolongation of pregnancy plus azithromycin for 5 days every month.

. The third group was the second test group in which the pregnant women administerated Azithromycin and clindamycin (Dalacin®) vaginal gel 5 times per month.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with <34 weeks of gestation,
* Hospitalization for risk of preterm labour,
* Threat of preterm labour, or preterm labour itself.
* Threat of preterm labour and preterm labour will have to be diagnosis cited in the medical record by the physician.
* Women at risk of preterm labour must have one of the following conditions cited in their record: sludge, short cervix, cerclage, or bulging membranes

Exclusion Criteria:

* Patients were excluded from the current study in case of the use of antibiotics within 14 days before the admission (except for pericerclage prophylaxis, or streptococcus B prophylaxis), PPROM or fetal extraction required <37 weeks.

Ages: 18 Years to 32 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Female above 18 years old
Study Population: Randomized Controlled prospective study
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Effect of Azithromycin in preventing premature labour | 6 monthes
  Main outcome was the number of days between diagnosis and composite event, defined as delivery or rupture of membranes or 2nd intervention aimed at prolonging pregnancy (such as cerclage or tocolysis) or censure (maternal death or transfer). The three groups were compared regarding this number of days

CONTACTS AND LOCATIONS:
Overall Officials: Raghda R.S Hussein, Principal Investigator — Beni-Suef University
Locations (1):
- Beni-Suef University teaching Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Pregnant women with risk for pre mature labour will adiminster azithromycin as monotherapy or polytherapy with clindamycin vaginal cream ,The efficacy of Azithromycin in preventing premature mature labour will be assessed